CLINICAL TRIAL: NCT03508050
Title: Clamping the Double Lumen Tube : A Novel Technique to Optimize One-Lung Ventilation
Brief Title: Clamping the Double Lumen Tube
Acronym: C-TDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Bussières (Other)
Responsible Party: Sponsor-Investigator, Jean Bussières, Anesthesiologist, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21436
Record Dates: First submitted 2017-09-27; First posted 2018-04-25 (Actual); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: One-lung Ventilation

STUDY DESIGN:
Intervention Model Description: Just before induction of anesthesia and according to the computerized randomization list generated by the statistical department, each of the 30 patients is allocated to one of the following groups:
  Control group : OLV with the specific lumen of the NVL opened to ambient air. Experimental group : OLV with a clamp on the specific lumen of the NVL
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamping double lumen tube (Experimental): Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
  Interventions: Device: Clamping the Double Lumen Tube
- Not Clamping double lumen tube (No Intervention): Not Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation

INTERVENTIONS:
Device: Clamping the Double Lumen Tube — Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
  Arms: Clamping double lumen tube

SUMMARY:
Nowadays, lung isolation techniques are an essential part of thoracic anesthesia. The two principal devices used in order to achieve one-lung ventilation (OLV) are the double lumen tube (DLT) and the bronchial blocker (BB). Even though DLT and BB have always been considered equally effective in lung isolation, a study recently published by Bussières et al. demonstrated the clear superiority of BB over DLT in terms of rapidity and quality of lung collapse. In order to explain this result, a physiologic study was recently conducted. During this project, some interesting discoveries were made. In fact, during lung isolation, while the chest is closed, there is a buildup of negative pressure in the NVL until pleural opening. Moreover, an absorption of ambient air through the lumen of the DLT or through the internal channel of the BB is observed. Putting all these elements together, a possible explanation for the superiority of BB over DLT was obtained. Indeed, in the first study of Bussières, the internal channel of BB was occluded. By doing so, there were no possible aspiration of ambient air in the NVL. This condition may have accelerated the absorption atelectasis of the NVL that occurs during lung collapse by reducing NVL volume and by conserving a higher alveolar partial pressure of oxygen in it.

The hypothesis is that when using a DLT in OLV, occluding the non-ventilated lung (NVL) lumen will reproduce the BB physiology by accelerating the second phase of lung deflation and giving a better quality of lung collapse compared to usual practice of keeping the non-ventilated lung opened to ambient air.

The main objective is to compare the speed and quality of complete lung deflation occurring during OLV with a DLT when the non-ventilated DLT lumen is occluded vs not occluded.

This randomized study will include a total of 30 patients scheduled for lung resection using video-assisted thoracoscopic surgery (VATS). Fifteen patients will compose the experimental group (NVL lumen occluded) and 15 other patients will be part of the control group (NVL lumen opened to ambient air).

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is a major consideration in thoracic anesthesia. Lung isolation, through the use of double-lumen tube (DLT) or bronchial blocker (BB), offers to the surgeon the intra-thoracic access he needs for the surgery. With the use of a DLT, the non-ventilated lung is isolated by disconnecting its specific lumen from the ventilator and keeping it opened to ambient air. With a BB, the BB cuff is inflated in the bronchus after a brief apnea period. Thereafter, only the dependent lung is ventilated.

Until recently, studies evaluating the quality of lung collapse with the use of DLT versus BB showed contradicting results and were not conclusive. However, in 2016, Bussières' research group obtained a faster lung collapse with the use of a BB with its internal channel occluded and a second period of apnea at pleural opening.

A review of the literature could not explain in details these results. In the 2000s, lung collapse during OLV was described as undergoing two distinct phases; the first phase occuring at the opening of the pleural cavity and corresponding to a quick but partial collapse secondary to the elastic recoil of the lung. The second phase, a slower one, being the reabsorption, by the vascular capillary bed, of the gas contained into the alveoli; the speed of this second phase being directly proportional to the solubility coefficient of the gas.

Since no previous studies had explanation for Bussières' unexpected results, they conducted a physiologic study to extensively determine the physiology of the non-ventilated lung (NVL) during OLV with the use of DLT and BB. Their results demonstrated that during lung isolation, while the chest is closed, there is a buildup of negative pressure in the NVL until pleural opening, when the lumen of the DLT or the internal channel of the BB are occluded. This phenomenon was observed for both lung isolation devices (BB and DLT). They also observed an absorption of ambient air through the lumen of the DLT and the internal channel of the BB when the lumen of both device was open to ambient air. These results probably explain why Bussières obtained a faster lung collapse with BB in their study. By occluding the internal channel of the BB they prevented the aspiration of ambient air in the NVL. This condition may have accelerated the absorption atelectasis of the NVL that occurs during the second phase of lung collapse by obtaining an initial lower lung volume containing a higher alveolar partial pressure of oxygen (PAO2) in the BB group.

Since these recent findings demonstrate that both lung isolation devices cause negative pressure and an aspiration of ambient air, it is possible that the occlusion of the specific lumen of the NVL of a DLT could reproduce the physiology of the lung isolation obtained with a BB with its internal channel occluded.

The hypothesis is that by withholding gas exchange between the NVL and ambient air from the beginning of OLV to the pleural opening, the resorption atelectasis will be facilitated. Consequently, lung collapse of the NVL will occur faster when clamping its specific lumen on the DLT instead of letting it communicate with ambient air like anesthesiologists usually do.

ELIGIBILITY:
Inclusion Criteria:

* Elective lung resection (lobectomies and segmentectomies) by VATS requiring OLV.
* More than 18 years old.
* Having read, understand and signed the consent form presented at the pre-operative evaluation

Exclusion criteria :

A- Pre-operative

1. Known or anticipated difficult tracheal intubation.
2. Bronchoscopic or CT-scan findings contraindicating the insertion of a DLT.
3. Severe COPD or asthma (FEV1 <50%).
4. Prior intrathoracic surgery (including cardiac surgeries).
5. Pleural or interstitial pathology.
6. Previous chemotherapy or thoracic radiotherapy.
7. Acute or chronic pulmonary infection.
8. Endobronchial mass.
9. Tracheostomy.

B- Post-randomisation

1. Bronchoscopic findings contraindicating the insertion of DLT.
2. VATS findings that cancel the surgery.
3. Severe desaturation (SatO2 < 90%) during the observation period.
4. Any need to reinflate the collapse lung.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Pelletier, MD, Principal Investigator — Laval University; Jean S Bussières, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Clayton-Smith A, Bennett K, Alston RP, Adams G, Brown G, Hawthorne T, Hu M, Sinclair A, Tan J. A Comparison of the Efficacy and Adverse Effects of Double-Lumen Endobronchial Tubes and Bronchial Blockers in Thoracic Surgery: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):955-66. doi: 10.1053/j.jvca.2014.11.017. Epub 2014 Dec 2. PMID 25753765
- [Background] Campos JH, Reasoner DK, Moyers JR. Comparison of a modified double-lumen endotracheal tube with a single-lumen tube with enclosed bronchial blocker. Anesth Analg. 1996 Dec;83(6):1268-72. doi: 10.1097/00000539-199612000-00024. PMID 8942598
- [Background] Bussieres JS, Somma J, Del Castillo JL, Lemieux J, Conti M, Ugalde PA, Gagne N, Lacasse Y. Bronchial blocker versus left double-lumen endotracheal tube in video-assisted thoracoscopic surgery: a randomized-controlled trial examining time and quality of lung deflation. Can J Anaesth. 2016 Jul;63(7):818-27. doi: 10.1007/s12630-016-0657-3. Epub 2016 May 2. PMID 27138896
- [Background] Pfitzner J, Peacock MJ, McAleer PT. Gas movement in the nonventilated lung at the onset of single-lung ventilation for video-assisted thoracoscopy. Anaesthesia. 1999 May;54(5):437-43. doi: 10.1046/j.1365-2044.1999.00845.x. PMID 10995140
- [Background] Joyce CJ, Baker AB, Kennedy RR. Gas uptake from an unventilated area of lung: computer model of absorption atelectasis. J Appl Physiol (1985). 1993 Mar;74(3):1107-16. doi: 10.1152/jappl.1993.74.3.1107. PMID 8482648
- [Background] Bardoczky GI, Engelman E, d'Hollander A. Continuous spirometry: an aid to monitoring ventilation during operation. Br J Anaesth. 1993 Nov;71(5):747-51. doi: 10.1093/bja/71.5.747. PMID 8251293
- [Background] Bussieres JS, Slinger P. Correct positioning of double-lumen tubes. Can J Anaesth. 2012 May;59(5):431-6. doi: 10.1007/s12630-012-9689-5. Epub 2012 Mar 7. No abstract available. English, French. PMID 22395826
- [Derived] Somma J, Couture EJ, Pelletier S, Provencher S, Moreault O, Lohser J, Ugalde PA, Vigneault L, Lemieux J, Somma A, Guay SE, Bussieres JS. Non-ventilated lung deflation during one-lung ventilation with a double-lumen endotracheal tube: a randomized-controlled trial of occluding the non-ventilated endobronchial lumen before pleural opening. Can J Anaesth. 2021 Jun;68(6):801-811. doi: 10.1007/s12630-021-01957-9. Epub 2021 Apr 2. PMID 33797018

RESULTS

PARTICIPANT FLOW:
Groups:
- Double Lumen Tube Clamp: Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
  Clamping the Double Lumen Tube: Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
- Control: Not Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
Period: Overall Study
Arm/Group | Double Lumen Tube Clamp | Control
Started | 20 | 17
Completed | 15 | 15
Not Completed | 5 | 2
Not completed — Pleural adhesions | 1 | 0
Not completed — Mucus plug | 1 | 0
Not completed — Negative biopsy, surgery cancelled | 3 | 1
Not completed — Sustained desaturation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
  Clamping the Double Lumen Tube: Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.67 (9.6) | 66.60 (6.5) | 65.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 30
Height (meter) [Mean (Standard Deviation); unit: meter] | 1.64 (0.10) | 1.62 (0.08) | 1.62 (0.09)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 67.73 (17.96) | 74.4 (14.88) | 71.07 (16.56)
Ideal body weight (kg) [Mean (Standard Deviation); unit: kg] | 59.27 (7.31) | 57.6 (6.25) | 58.43 (6.74)
Forced Expiratory Volume - 1 sec (FEV1) [Mean (Standard Deviation); unit: % predicted value] | 93.27 (15.29) | 96.27 (16.1) | 94.77 (15.5)
Tiffeneau index (FEV1/FVC ratio) [Mean (Standard Deviation); unit: ratio of predicted value] | 71.93 (10.29) | 73.33 (6.4) | 72.63 (8.45)

OUTCOME MEASURES:

1. Primary Outcome: T50-3
Description: Moment where the probability of having a complete lung collapse is 50%
Time Frame: From the beginning of surgery (pleural opening) until 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 14 | 15
minutes
  First random videoclip analysis | 31.87 (3.68) | 63.81 (10.77)
  Second random videoclip analysis | 33.30 (3.71) | 60.82 (7.51)

2. Secondary Outcome: Complete Lung Collapse (CLC-clinical)
Description: The time required to obtain CLC. This end-point is assessed clinically by the surgeon during the surgery
Time Frame: From the beginning of surgery (pleural opening) until 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Double Lumen Tube Clamp: Clamping the non-dependent lung's lumen of the double lumen tube during closed chest one-lung ventilation
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
minutes | 28.67 (15.04) | 59.47 (20.79)

3. Secondary Outcome: O2 Concentration of Expired Air at Pleural Opening
Description: A measure of the O2 concentration of the expiratory air at pleural opening
Time Frame: From pleural opening and lasting 60 seconds
Measure: Mean (Standard Deviation); unit: % of oxygen
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
% of oxygen | 41.87 (18.61) | 11.93 (3.65)

4. Secondary Outcome: Expiratory Volume at Pleural Opening
Description: A measure of the expiratory volume (EV) at pleural opening
Time Frame: From pleural opening and lasting 60 seconds
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
ml | 178.53 (138.12) | 421.13 (199.9)

5. Secondary Outcome: O2 Concentration of Expired Air at the Beginning of One-lung Ventilation
Description: A measure of the O2 concentration of the expiratory air at the beginning of one-lung ventilation (OLV)
Time Frame: From the beginning of one-lung ventilation and lasting 60 seconds
Measure: Mean (Standard Deviation); unit: % of oxygen
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
% of oxygen | 40.93 (5.87) | 35.13 (3.89)

6. Secondary Outcome: Optimization of Lung Collapse
Description: Number of Participants needing Other Interventions to Optimize Lung Collapse
Time Frame: From the beginning of surgery (pleural opening) until 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
Participants | 0 | 1

7. Secondary Outcome: Quality of Oxygenation During One-lung Ventilation (PaO2 )
Description: An evaluation of the PaO2 during one-lung ventilation
Time Frame: 25 minutes after pleural opening
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 14
mmHg | 162.86 (68.71) | 128.60 (57.69)

8. Secondary Outcome: Quality of Oxygenation During One-lung Ventilation (SaO2)
Description: An evaluation of the SaO2during one-lung ventilation
Time Frame: 25 minutes after pleural opening
Measure: Mean (Standard Deviation); unit: % of oxygen saturation
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 14 | 15
% of oxygen saturation | 97.78 (1.79) | 95.67 (2.09)

9. Secondary Outcome: Surgery Duration
Description: Time required for completion of the surgery
Time Frame: From the beginning of surgery (pleural opening) until 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
minutes | 89.27 (34.01) | 88.40 (30.39)

10. Secondary Outcome: Postoperative Atelectasis
Description: Number of atelectasis detected by Postoperative X-Ray
Time Frame: End of hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
Participants | 1 | 6

11. Secondary Outcome: Quality of Lung Collapse (Clinical) at 0 Minute
Description: A clinical evaluation, by the thoracic surgeon, of the quality of the surgical exposure following lung collapse using a visual scale graduated from 1 to 3. Score 1 = No lung collapse, Score 2 = Partial lung collapse, Score 3 = Complete lung collapse Scale title: Visual grading scale of lung collapse Higher score means a better outcome
Time Frame: At pleural opening (0 minute)
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
Participants
  No lung collapse | 0 | 1
  Partial lung collapse | 14 | 14
  Complete lung collapse | 1 | 0

12. Secondary Outcome: Quality of Lung Collapse (Clinical) at 10 Minutes
Description: as for outcome 11
Time Frame: 10 minutes after pleural opening
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
Participants
  No lung collapse | 1 | 0
  Partial lung collapse | 14 | 14
  Complete lung collapse | 0 | 1

13. Secondary Outcome: Quality of Lung Collapse (Clinical) at 20 Minutes
Description: as for outcome 11
Time Frame: 20 minutes after pleural opening
Measure: Count of Participants; unit: Participants
Arm/Group | Double Lumen Tube Clamp | Control
Number analyzed (Participants) | 15 | 15
Participants
  No lung collapse | 0 | 0
  Partial lung collapse | 8 | 14
  Complete lung collapse | 7 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of the surgery through completion of surgery. Moreover, the first PACU thoracic x-ray of each patient was analyzed by a radiologist in order to detect anomalies.
Arm/Group | Double Lumen Tube Clamp | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/17
Other Adverse Events (participants affected / at risk) | 1/15 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Lumen Tube Clamp (N=20) | Control (N=17)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Sustained desaturation under 90% of SaO2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.06% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Lumen Tube Clamp (N=15) | Control (N=15)
X-ray anomalies (Respiratory, thoracic and mediastinal disorders) | 1 | 7 — Post-operative thoracic x-ray anomalies

LIMITATIONS AND CAVEATS:
Post-randomisation exclusions. Most of them due to negative biopsies cancelling the need of a lobectomy/segmentectomy.

The study was single blinded. (the anesthesiologist knew in which group the patient was but the surgeon was blinded)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03508050/Prot_SAP_000.pdf